CLINICAL TRIAL: NCT02067273
Title: Transcranial Magnetic Stimulation for CRPS
Brief Title: Transcranial Magnetic Stimulation (TMS) for CRPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Chief, Division of Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25894-2
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Transcranial Magnetic Stimulation

ARMS (2):
- TMS Intervention for 5 days (Experimental): Application of Transcranial Magnetic Stimulation (TMS) for up to 5 days
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS Intervention for 1 day (Experimental): Application of Transcranial Magnetic Stimulation (TMS) for 1 day
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS)

SUMMARY:
The purpose of this pilot study is to test the durability of response to Transcranial Magnetic Stimulation (TMS) for the symptoms of Complex Regional Pain Syndrome (CRPS). The investigators will test various methods of TMS for varying lengths of time in a pilot study to investigate what the clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of CRPS (complex regional pain syndrome)
* Average pain level reported on Numerical Rating Scale meets entry criteria
* Ability to perform the experimental task and procedures.

Exclusion Criteria:

* MRI contraindication (metal implants or devices, claustrophobia)
* TMS Contraindication (eg metal implant or devices near the site of stimulation)
* History of epilepsy
* History of a psychological or psychiatric disorder that would interfere with study procedures, at the discretion of the researcher.
* Neurologic illness that would interfere with brain integrity
* Current medical condition or medication use that would interfere with study procedures or data integrity, at the discretion of the researcher.
* Currently pregnant or planning to become pregnant.
* On going legal action or disability claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

REFERENCES:
- See also: Related Info — http://snapl.stanford.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Intervention for 1 Day: Application of Transcranial Magnetic Stimulation (TMS) for 1 day
  Transcranial Magnetic Stimulation (TMS)
- TMS Intervention for 5 Days: Application of Transcranial Magnetic Stimulation (TMS) once a day for 5 days
  Transcranial Magnetic Stimulation (TMS)
Period: Overall Study
Arm/Group | TMS Intervention for 1 Day | TMS Intervention for 5 Days
Started | 5 | 15
Completed | 5 | 12
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMS Intervention for 1 Day | TMS Intervention for 5 Days | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Categorical [Count of Participants; unit: Participants] — Population: Only data from participants who completed the study were analyzed.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 4 | 11 | 15
    >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Only data from participants who completed the study were analyzed.
  years | 49.8 (16.47) | 42.92 (13.69) | 44.94 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Present Pain Intensity
Description: Present pain intensity was reported by participants using a visual analog scale (VAS) from scores ranging from 1-10; lower scores represent less pain, higher scores represent more severe pain.
Time Frame: Baseline, post-treatment, one week follow-up
Population: Data from participants who completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- TMS Intervention (1 Day): Application of Transcranial Magnetic Stimulation (TMS) for 1 day
  Transcranial Magnetic Stimulation (TMS)
- TMS Intervention (5 Days): Application of Transcranial Magnetic Stimulation (TMS) once a day for 5 days
  Transcranial Magnetic Stimulation (TMS)
Arm/Group | TMS Intervention (1 Day) | TMS Intervention (5 Days)
Number analyzed (Participants) | 5 | 12
Units on a scale
  Baseline | 6.5 (2.3) | 6.3 (1.4)
  Post-treatment | 3.1 (3.1) | 3.7 (3.0)
  One week follow-up | 4.6 (4.0) | 4.3 (2.7)

ADVERSE EVENTS:
Arm/Group | TMS Intervention for 1 Day | TMS Intervention for 5 Days
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 1/5 | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Intervention for 1 Day (N=5) | TMS Intervention for 5 Days (N=15)
Headache (General disorders) | 1 (1) | 7 (7)
Muscle spasms (General disorders) | 0 | 2 (2)
Procedural discomfort (General disorders) | 0 | 1 (1)
Increased pain (General disorders) | 0 | 2 (2)
Neck pain (General disorders) | 0 | 2 (2)
Nausea (General disorders) | 0 | 1 (1)
Gingival pain (General disorders) | 0 | 1 (1)
Fatigue (General disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes